CLINICAL TRIAL: NCT02578706
Title: Targeting Platelets in Chronic HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Meagan O'Brien, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 14-1374; R56HL127995-01 (NIH)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: HIV-1 Infection
Keywords: HIV; Aspirin; Clopidogrel; Platelet; Inflammation; Cardiovascular disease; Arachidonic acid; Cyclooxygenase inhibitor; ADP inhibitor; Immune activation; Monocyte; Coagulation; Thrombogenicity
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases; Thrombosis | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aspirin and placebo (Active Comparator): At week 0, participants will be administered aspirin 81mg (one tablet) and placebo for clopidogrel 75 mg (one tablet) once daily. At week 24, participants will stop both study product tablets.
  Interventions: Drug: Aspirin; Drug: Placebo
- Clopidogrel and placebo (Active Comparator): At week 0, participants will be administered clopidogrel 75 mg (one tablet) and placebo for aspirin 81 mg (one tablet) once daily. At week 24, participants will stop both study product tablets.
  Interventions: Drug: Clopidogrel; Drug: Placebo
- Placebos only (Placebo Comparator): At week 0, participants will be administered placebo for aspirin 81 mg (one tablet) and placebo for clopidogrel 75mg (one tablet) once daily. At week 24, participants will stop both study product tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75mg
  Other Names: Plavix
  Arms: Clopidogrel and placebo
Drug: Aspirin — 81 mg
  Arms: Aspirin and placebo
Drug: Placebo

SUMMARY:
Advances in antiretroviral therapy (ART) have resulted in increased survival of the HIV-infected population; however, this gain in longevity is associated with an increased risk of cardiovascular disease (CVD). Although ART and traditional risk factors contribute to CVD in this population, heightened markers of immune activation, inflammation, and coagulation independently predict morbidity and mortality, suggesting that dysregulation of these systems plays a significant role in the increased risk of CVD. The investigators believe that platelet activation is an important driver in HIV-associated immune activation, inflammation, and coagulation, leading to an increased CVD pathophysiology and risk. Platelets initiate thrombus formation and also play a key role in vascular inflammation by releasing pro-inflammatory mediators and cross-talking with other relevant cell types including leukocytes. Researchers have described platelet hyperreactivity in chronic HIV infection. Importantly, the investigators demonstrated that one week of anti-platelet therapy (aspirin) decreased platelet activation and immune activation, with an improved trend in inflammation and immune parameters. The overall hypothesis is that platelet activation is a major driver of immune activation, inflammation, and thrombosis in ART-treated HIV infected patients. The purpose of the proposed proof-of-concept study is to understand the mechanism(s) by which anti-platelet therapy improves immune and inflammatory parameters in chronic HIV infection. To test this, the immune modulating and anti-inflammatory effects of 24 weeks of the anti-platelet drug aspirin as compared to the anti-platelet drug clopidogrel will be evaluated. Given their different mechanisms of action and inhibitory potency, the investigators can differentiate whether the potential benefits are mediated via inhibition of arachidonic acid (aspirin) or inhibition of ADP (clopidogrel) or by the antithrombotic activity. A secondary goal is to perform multidimensional assays of platelet activity and thrombogenicity alongside immune activation assays and careful assessments of traditional risk factors and medication regimens, to understand which parameters are highly associated with thrombogenicity.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial of 40 HIV-1 infected participants on stable ART randomized in a 1:1:1 ratio to aspirin 81mg daily vs clopidogrel 75mg daily vs placebo for 24 weeks. A subset of patients in each arm will participate in a sub-study to evaluate thrombogenicity, to be performed prior to the first study treatment and at 24 weeks of study treatment. 10 HIV uninfected control subjects will participate the study to evaluate baseline characteristics.

The primary endpoint is to determine the impact of aspirin as compared to clopidogrel on immune activation and inflammation in HIV infected, ART treated adults. This will be determined by measuring the change in the clinically relevant soluble marker of inflammation sCD14 over 24 weeks of study drug. Secondary objectives will be to measure safety and tolerability, to measure the effects of study drugs on important soluble markers of inflammation (sCD163, IL-6, d-dimer, sTNFRI and II), by measuring monocyte subsets (CD14, CD16, CD69), by measuring platelet activation by light transmission aggregometry, monocyte-platelet aggregates, and soluble CD40L, by measuring clot formation kinetics by thromboelastography, and in a subset of patients, by measuring thrombogenicity by Badimon Chamber and cholesterol uptake by monocytes.

ELIGIBILITY:
HIV infected participants:

Inclusion Criteria:

* HIV-1 infection
* Currently on continuous ART for ≥48 weeks prior to study entry. NOTE: This is defined as continuous active therapy with no treatment interruption longer than 7 consecutive days and a total duration off-treatment of no more than 14 days during the 48 weeks prior to entry.
* No change in ART regimen within the 12 weeks prior to study entry (except as noted below).

NOTE: Modifications of ART dosing during the 12 weeks prior to entry are permitted. In addition, the change in formulation (eg, from standard formulation to fixed dose combination or single tablet regimen) or dosing (eg, from once a day to twice a day) is allowed within 12 weeks prior to entry. Within-class single drug substitution (eg, switch from nevirapine to efavirenz or from atazanavir to darunavir), are not allowed within 12 weeks prior to entry. No other changes in ART in the 12 weeks prior to entry are permitted.

* Screening HIV-1 RNA must be <50 copies/mL and performed by any FDA-approved assay at any US laboratory that has a CLIA certification or its equivalent within 45 days prior to study entry.
* Maintain ART-mediated viral suppression for at least 48 weeks prior to study entry defined as:

A. At least one HIV-1 RNA test result obtained at any time point greater than 48 weeks prior to study entry must be BLQ and must be performed by any FDA-approved assay at a CLIA-certified laboratory.

AND B. All HIV-1 RNA tests reported during the 48 weeks prior to study entry must be BLQ and must be performed by any FDA-approved assay at a CLIA-certified laboratory.

NOTE: A single RNA "blip" of ≤500 copies/mL is permissible if RNA levels most recent before and after (may include the screening HIV-1 RNA test) are BLQ for the assay.

* The following laboratory values obtained within 45 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent.

  * Absolute neutrophil count (ANC) ≥750/mm3
  * Hemoglobin ≥9.0 g/dL for female subjects and ≥10.0 g/dL for male subjects
  * Platelet count >100,000/mm3
  * Prothrombin time (PT) <1.2 x upper limit normal (ULN)
  * Partial thromboplastin time (PTT) <1.5 x ULN
  * Calculated creatinine clearance (CrCl) ≥30 mL/min, as estimated by the Cockroft-Gault formula
  * Aspartate aminotransferase (AST) (SGOT) ≤2 x ULN.
  * Alanine aminotransferase (ALT) (SGPT) ≤2 x ULN.
  * Alkaline phosphatase ≤2 x ULN.
  * Total bilirubin ≤2.5 x ULN. If the subject if taking an indinavir- or atazanavir-containing regimen at the time of screening, a total bilirubin of ≤5 x ULN is acceptable.
* Female study volunteers of reproductive potential (pre-menopausal women who have not had a sterilization procedure (eg, hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy)) must have a negative serum or urine pregnancy test performed within 24 hours before initiating the protocol-specified medication(s) unless otherwise specified by product labeling. Women are considered menopausal if they have not had a menses for at least 12 months and have a FSH (follicle stimulating hormone) of greater than 40 IU/L or, if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

If the female volunteer is not of reproductive potential (women who are menopausal, defined as not having had a menses for at least 12 months with an FSH of greater than 40 IU/L, or if FSH testing is not available, have had amenorrhea for 24 consecutive months, or women who have undergone surgical sterilization, (eg, hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy)), she is eligible without requiring the use of a contraceptive method. Acceptable documentation of sterilization is subject reported history of hysterectomy, bilateral oophorectomy, tubal ligation, tubal micro-insert, menopause, or the partner with vasectomy/azoospermia.

* If participating in sexual activity that could lead to pregnancy, the female study volunteer must be willing to use contraception while receiving protocol-specified medication(s) and for the washout period of 4 weeks. At least one of the following methods MUST be used:

  * Condoms (male or female), with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive As hormone-based contraceptives (oral, transdermal, or subdermal) can affect coagulopathy biomarkers, subjects who plan on using such a contraceptive during the study must be taking the same product for ≥4 weeks prior to screening and be encouraged to continue throughout the duration of the study, if medically feasible.
* No documented opportunistic infections within 24 weeks prior to study entry
* Karnofsky performance score >70 within 45 days prior to study entry
* Ability and willingness of subject or legal guardian/representative to provide written informed consent.
* Willingness to refrain from the use of aspirin or any aspirin-related product (other than the study drug), including NSAIDs, from time of screening visit through the end of the 24 week trial.

NOTE: Acetaminophen-based products may be used before and during the trial when analgesics are required.

Exclusion Criteria:

• Current malignancy (except non-melanoma cancer of the skin not requiring systemic chemotherapy or radiation therapy).

NOTE: Carcinoma in situ of the cervix or anus is not considered exclusionary.

* Prior history of malignancy if the subject is not disease free for 24 or more weeks prior to study entry.
* Current use of non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin that cannot be interrupted for clinical reasons. Examples of clinical reasons include, but are not limited to, known and documented cardiovascular disease (history of MI, coronary artery bypass graft surgery, percutaneous coronary intervention, stroke, transient ischemic attack, peripheral arterial disease with ABI <0.9 or claudication).
* Current diagnosis of diabetes with HbA1c ≥8% at screening.
* Use of lipid-lowering medications including: statins, fibrates, niacin (dose ≥250 mg daily), and fish-oil/omega 3 fatty acids (dose >1000 mg of marine oils daily).
* Known cirrhosis
* Known chronic active hepatitis B NOTE: Active hepatitis B is defined as hepatitis B surface antigen positive and hepatitis B DNA positive within 24 weeks prior to study entry; subjects with hepatitis B virus (HBV) DNA BLQ for greater than 24 weeks prior to study entry are eligible.
* Known chronic active hepatitis C NOTE: Active hepatitis C is defined as a detectable plasma HCV RNA level within 24 weeks prior to study entry; subjects with HCV RNA BLQ for greater than 24 weeks prior to study entry are eligible.
* Known inflammatory conditions, such as, but not limited to, rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), sarcoidosis, inflammatory bowel disease (IBD), chronic pancreatitis, autoimmune hepatitis, Adult Stills disease, Rheumatic heart disease, bursitis.
* Breastfeeding or pregnant
* Previous intolerance or allergy to aspirin or any aspirin products or clopidogrel.
* Frequent use of aspirin or aspirin products (NSAIDs), defined as an average of 2 or more times per week in the last 12 weeks prior to study entry.
* Immunosuppressant use, such as, but not limited to, systemic or potentially systemic glucocorticoids (including injected, ie, intra-articular, nasal or inhaled steroids), azathioprine, tacrolimus, mycophenolate, sirolimus, rapamycin, methotrexate, or cyclosporine within 45 days prior to study entry.
* Use of any systemic antineoplastic or immunomodulatory treatment, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry.

NOTE: Routine standard of care, including hepatitis A and/or B, human papilloma virus, influenza, pneumococcal, and tetanus vaccines are permitted if administered at least 7 days before study entry and before biomarker/peripheral blood mononuclear cell (PBMC) blood collections.

* Heavy alcohol use as defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA)
* Alcohol or drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Current use of anticoagulation therapy or conditions requiring use of anticoagulants, use such as, but not limited to warfarin (Coumadin), rivaroxaban (Xarelto), clopidogrel (Plavix), dabigatran (Pradaxa), apixaban (Eliquis), heparin, ticlopidine (Ticlid), Presugrel (Effient).
* History of coagulopathy, deep venous thrombosis, pulmonary embolism.
* Known active or recent (not fully resolved within 4 weeks prior to study entry) invasive bacterial, fungal, parasitic, or viral infections.

NOTE: Recurrent herpes simplex virus (HSV) is not exclusionary. Subjects on antiviral prophylaxis for HSV or VZV are encouraged to remain on treatment for the duration of the study if medically feasible.

* Serious illness or trauma requiring systemic treatment and/or hospitalization within 4 weeks prior to study entry.
* History of bleeding conditions such as peptic ulcer disease, hemophilia, von Willebrand disease, idiopathic thrombocytopenic purpura.
* History of thrombotic disorders such as protein C or S deficiency.
* History of gastrointestinal (GI) bleeding within the past 6 months prior to study entry.
* History of intracranial hemorrhage.

HIV-uninfected participants:

Inclusion criteria:

• HIV uninfected

Exclusion criteria:

• Current malignancy (except non-melanoma cancer of the skin not requiring systemic chemotherapy or radiation therapy).

NOTE: Carcinoma in situ of the cervix or anus is not considered exclusionary.

* Prior history of malignancy if the subject is not disease free for 24 or more weeks prior to study entry.
* Current use of non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin that cannot be interrupted for clinical reasons.
* Current diagnosis of diabetes with HbA1c ≥8% at screening.
* Use of lipid-lowering medications including: statins, fibrates, niacin (dose ≥250 mg daily), and fish-oil/omega 3 fatty acids (dose >1000 mg of marine oils daily).
* Known cirrhosis
* Known chronic active hepatitis B
* Known chronic active hepatitis C
* Known inflammatory conditions, such as, but not limited to, rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), sarcoidosis, inflammatory bowel disease (IBD), chronic pancreatitis, autoimmune hepatitis, Adult Stills disease, Rheumatic heart disease, bursitis.
* Breastfeeding or pregnant
* Previous intolerance or allergy to aspirin or any aspirin products or clopidogrel.
* Frequent use of aspirin or aspirin products (NSAIDs), defined as an average of 2 or more times per week in the last 12 weeks prior to study entry.
* Immunosuppressant use, such as, but not limited to, systemic or potentially systemic glucocorticoids (including injected, ie, intra-articular, nasal or inhaled steroids), azathioprine, tacrolimus, mycophenolate, sirolimus, rapamycin, methotrexate, or cyclosporine within 45 days prior to study entry.
* Use of any systemic antineoplastic or immunomodulatory treatment, investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry.

NOTE: Routine standard of care, including hepatitis A and/or B, human papilloma virus, influenza, pneumococcal, and tetanus vaccines are permitted if administered at least 7 days before study entry and before biomarker/peripheral blood mononuclear cell (PBMC) blood collections.

* Heavy alcohol use as defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA)
* Alcohol or drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Current use of anticoagulation therapy or conditions requiring use of anticoagulants, use such as, but not limited to warfarin (Coumadin), rivaroxaban (Xarelto), clopidogrel (Plavix), dabigatran (Pradaxa), apixaban (Eliquis), heparin, ticlopidine (Ticlid), Presugrel (Effient).
* History of coagulopathy, deep venous thrombosis, pulmonary embolism.
* Known active or recent (not fully resolved within 4 weeks prior to study entry) invasive bacterial, fungal, parasitic, or viral infections.

NOTE: Recurrent herpes simplex virus (HSV) is not exclusionary. Subjects on antiviral prophylaxis for HSV or VZV are encouraged to remain on treatment for the duration of the study if medically feasible.

* Serious illness or trauma requiring systemic treatment and/or hospitalization within 4 weeks prior to study entry.
* History of bleeding conditions such as peptic ulcer disease, hemophilia, von Willebrand disease, idiopathic thrombocytopenic purpura.
* History of thrombotic disorders such as protein C or S deficiency.
* History of gastrointestinal (GI) bleeding within the past 6 months prior to study entry.
* History of intracranial hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meagan O'Brien, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Juan Badimon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] O'Brien M, Montenont E, Hu L, Nardi MA, Valdes V, Merolla M, Gettenberg G, Cavanagh K, Aberg JA, Bhardwaj N, Berger JS. Aspirin attenuates platelet activation and immune activation in HIV-1-infected subjects on antiretroviral therapy: a pilot study. J Acquir Immune Defic Syndr. 2013 Jul 1;63(3):280-8. doi: 10.1097/QAI.0b013e31828a292c. PMID 23406976
- [Background] Miller EA, Gopal R, Valdes V, Berger JS, Bhardwaj N, O'Brien MP. Soluble CD40 ligand contributes to dendritic cell-mediated T-cell dysfunction in HIV-1 infection. AIDS. 2015 Jul 17;29(11):1287-96. doi: 10.1097/QAD.0000000000000698. PMID 26091297
- [Background] Viswanathan GN, Marshall SM, Balasubramaniam K, Badimon JJ, Zaman AG. Differences in thrombus structure and kinetics in patients with type 2 diabetes mellitus after non ST elevation acute coronary syndrome. Thromb Res. 2014 May;133(5):880-5. doi: 10.1016/j.thromres.2014.01.033. Epub 2014 Feb 1. PMID 24582462
- [Background] Hutter R, Speidl WS, Valdiviezo C, Sauter B, Corti R, Fuster V, Badimon JJ. Macrophages transmit potent proangiogenic effects of oxLDL in vitro and in vivo involving HIF-1alpha activation: a novel aspect of angiogenesis in atherosclerosis. J Cardiovasc Transl Res. 2013 Aug;6(4):558-69. doi: 10.1007/s12265-013-9469-9. Epub 2013 May 10. PMID 23661177
- [Background] Arazi HC, Badimon JJ. Anti-inflammatory effects of anti-platelet treatment in atherosclerosis. Curr Pharm Des. 2012;18(28):4311-25. doi: 10.2174/138161212802481264. PMID 22236116

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Only: At week 0, participants will be administered placebo for aspirin 81 mg (one tablet) and placebo for clopidogrel 75mg (one tablet) once daily. At week 24, participants will stop both study product tablets.
Period: Overall Study
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Started | 9 | 10 | 8
Completed | 8 | 5 | 8
Not Completed | 1 | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only | Total
Number analyzed (Participants) | 9 | 10 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.9) | 44.2 (8.3) | 50.75 (11.7) | 46.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 4 | 17
  Male | 2 | 4 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in sCD14 From Baseline to Week 24
Description: Soluble CD14 (sCD14) levels in blood. sCD14 is a nonspecific maker of monocyte activation.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
pg/mL | 35.75 (231.87) | -251.40 (201.33) | -101.75 (339.34)

2. Secondary Outcome: Number of Subjects With at Least One Grade 3 or Higher Sign/Symptom or Laboratory Abnormality
Description: Safety as measured by a Summary of the number of subjects with at least one grade 3 or higher sign/symptom or laboratory abnormality. A grade 3 sign/symptom was defined as medically significant but not immediately life threatening.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
Participants | 0 | 1 | 0

3. Secondary Outcome: Change in Classical Monocyte Subsets From Baseline to Week 24
Description: The classical monocyte is characterized by high level expression of the CD14 cell surface receptor (CD14++ CD16- monocyte)
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: 10^3 cells/µl
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
10^3 cells/µl | -0.09 (0.13) | -0.12 (0.19) | -0.04 (0.20)

4. Secondary Outcome: Change in Intermediate Monocyte Subsets From Baseline to Week 24.
Description: The intermediate monocyte with high level expression of CD14 and low level expression of CD16 (CD14++CD16+ monocytes).
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: 10^3 cells/µl
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
10^3 cells/µl | 0.02 (0.18) | 0.06 (0.19) | 0.04 (0.18)

5. Secondary Outcome: Change in Non-classical Monocyte Subsets From Baseline to Week 24
Description: The non-classical monocyte shows low level expression of CD14 and additional co-expression of the CD16 receptor (CD14+CD16++ monocyte).[
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: 10^3 cells/µl
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
10^3 cells/µl | 0.002 (0.04) | 0.03 (0.05) | -0.03 (0.11)

6. Secondary Outcome: Change in Monocyte Activation sCD163 From Baseline to Week 24
Description: Soluble CD163 is a specific macrophage activation marker, associated with morphological disease grade. A high sCD163 indicates more disease.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: 10^3 cells/µl
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
10^3 cells/µl | 26.88 (137.06) | 15.8 (102.24) | -63.38 (138.19)

7. Secondary Outcome: Change in IL-6 From Baseline to Week 24
Description: Interleukin 6 gene encodes a cytokine that functions in inflammation and implicated in a variety of inflammatory-associated disease states.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
pg/mL | -0.36 (1.01) | 0.02 (4.08) | 0.85 (2.61)

8. Secondary Outcome: Change in D-dimer From Baseline to Week 24
Description: D-Dimer level looks at coagulation of blood. D-dimers are not normally present in blood except when coagulation has occurred.
Time Frame: Baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
mcg/L | -295.99 (1898.66) | 151.96 (721.59) | 1109.38 (2664.77)

9. Secondary Outcome: Change in sTNFR I From Baseline to Week 24
Description: Soluble tumor necrosis factor receptor (sTNFR) serum concentration
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
pg/ml | 137.77 (262.09) | 59.46 (38.18) | 19.78 (98.66)

10. Secondary Outcome: Change in sTNFR II From Baseline to Week 24
Description: Soluble tumor necrosis factor receptor (sTNFR) serum concentration
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
pg/ml | 283.13 (444.62) | 347.00 (1103.85) | 4.25 (486.28)

11. Secondary Outcome: Change in sCD40L From Baseline to Week 24
Description: Soluble CD40-ligand levels
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
pg/mL | -28.05 (147.34) | -25.68 (188.83) | 13.65 (106.45)

12. Secondary Outcome: Change in Platelet Aggregometry in Response to ADP 20µM From Baseline to Week 24
Description: Change in % platelet aggregation in response to stimulation by Adenosine Diphosphate (ADP) from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % platelet aggregation
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
% platelet aggregation | -7.25 (8.06) | -32.40 (25.41) | -6.50 (10.61)

13. Secondary Outcome: Change in Platelet Aggregometry in Response to Collagen 2µg/mL From Baseline to Week 24
Description: Change in % platelet aggregation in response to stimulation by Collagen 2µg/mL from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % platelet aggregation
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
% platelet aggregation | -40.37 (26.70) | -9.60 (14.69) | 8.62 (21.20)

14. Secondary Outcome: Change in Platelet Aggregometry in Response to Epi 5µM From Baseline to Week 24
Description: Change in % platelet aggregation in response to stimulation by light transmission aggregometry as measured by epinephrine 5µM from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % platelet aggregation
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
% platelet aggregation | -35.25 (31.56) | -21.40 (42.02) | -10.63 (32.07)

15. Secondary Outcome: Change in Spontaneous Platelet Aggregometry From Baseline to Week 24
Description: Change in spontaneous % platelet from baseline to week 24. Spontaneous platelet aggregation?
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % platelet
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
% platelet | -0.75 (1.28) | -0.60 (2.19) | -0.88 (2.23)

16. Secondary Outcome: Change in Platelet Aggregometry in Response to Arachidonic Acid 1500µM From Baseline to Week 24
Description: Change in % platelet aggregation in response to stimulation by arachidonic acid 1500µM from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % platelet aggregation
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
% platelet aggregation | -53.33 (41.91) | -31.00 (0) | -13.25 (35.88)

17. Secondary Outcome: Change in Monocyte Platelet Aggregates From Baseline to 24 Weeks
Description: Change in % platelet monocyte aggregates from baseline to week 24
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % platelet monocyte aggregates
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
% platelet monocyte aggregates | 10.55 (16.41) | 3.88 (12.02) | 8.96 (24.59)

18. Secondary Outcome: Change in Coagulation Time (CT) From Baseline to 24 Weeks
Description: Clot formation kinetics, or coagulation time, is measured using thromboelastography. time to 2mm amplitude in seconds.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
seconds | 3.00 (23.30) | 1.00 (24.30) | -13.13 (33.75)

19. Secondary Outcome: Change in Clot Formation Time (CFT) From Baseline to 24 Weeks
Description: Clot formation time is measured using thromboelastography. time from 2 to 20 mm amplitude in seconds.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
seconds | -1.00 (7.58) | 2.00 (4.69) | 1.63 (15.62)

20. Secondary Outcome: Change in Maximum Clot Firmness (MCF) From Baseline to 24 Weeks
Description: Maximum Clot Firmness (MCF) is measured using thromboelastography. maximum ampliture in mm
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
mm | 1.38 (1.69) | 1.20 (2.77) | 0.38 (4.47)

21. Secondary Outcome: Change in Alpha Angle From Baseline to 24 Weeks
Description: Alpha angle is measured using thromboelastography, measured by a tangent to the clotting curve through the 2mm point
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
degree | 0.00 (1.85) | -0.60 (1.14) | -0.50 (3.25)

22. Secondary Outcome: Change in Thrombus Formation (Low Shear) From Baseline to 24 Weeks
Description: substudy - Change in thrombus formation by Badimon chamber (low shear) from baseline to 24 weeks. Thrombus formation on a blood vessel measured by immunohistochemistry staining of tissue cross sections. μ(2)/mm is the area of thrombus. The low shear chamber (inner lumen diameter 0.2 mm, Reynolds number 30, shear rate 500 s- 1) simulates flow conditions of a normal coronary artery.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: μ(2)/mm
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
μ(2)/mm | -1036 (1364.39) | -899.20 (708.83) | -203.75 (1741.07)

23. Secondary Outcome: Change in Thrombus Formation (High Shear) From Baseline to 24 Weeks
Description: substudy - Change in thrombus formation by Badimon chamber (high shear) from baseline to 24 weeks. Thrombus formation on a blood vessel measured by immunohistochemistry staining of tissue cross sections. The high shear chambers (inner lumen diameter 0.1 mm, Reynolds number 60, shear rate 1690 s- 1) mimic the rheologic conditions of a moderately stenosed coronary artery.
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: μ(2)/mm
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 8 | 5 | 8
μ(2)/mm | -3052.20 (2859.52) | -2798.80 (3416.15) | -753.00 (1983.83)

24. Secondary Outcome: Change in Cholesterol Uptake by Monocytes
Description: substudy
Time Frame: baseline and 24 weeks
Population: data not collected
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebo Only
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Aspirin and Placebo | Clopidogrel and Placebo | Placebos Only
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin and Placebo (N=9) | Clopidogrel and Placebo (N=10) | Placebos Only (N=8)
Cholecystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — not related to study drug

LIMITATIONS AND CAVEATS:
This study was powered assuming that 40 study participants would be assigned per arm, however less than 10 participants were assigned per arm, therefore more participants would be needed to observe significant differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes